CLINICAL TRIAL: NCT00002569
Title: Phase III Intergroup Randomized Comparison of Radiation Alone vs. Pre-Radiation Chemotherapy for Pure and Mixed Anaplastic Oligodendrogliomas
Brief Title: Radiation Therapy With or Without Chemotherapy in Treating Patients With Anaplastic Oligodendroglioma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); North Central Cancer Treatment Group (Network); SWOG Cancer Research Network (Network); Eastern Cooperative Oncology Group (Network); NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-9402; CDR0000063603; CAN-NCIC-CE2; E-R9402; NCCTG-927252; SWOG-9402; INT-0149
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult anaplastic oligodendroglioma; adult mixed glioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Oligodendroglioma; Glioma | interventions — Lomustine; Procarbazine; Vincristine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiation therapy (RT) alone (Active Comparator): Radiation therapy (RT) alone - External Beam RT 59.4 Gy (1.8 Gy x 33 fractions, 5 days a week) to MR defined tumor volume.
  Interventions: Radiation: radiation therapy
- Intensive pre-treatment chemotherapy and radiation therapy (Experimental): Intensive pre-treatment chemotherapy (Day 1 CCNU 130 mg/m2 p.o., Day 8 - Vincristine 1.4 mg/m2 i.v., Days 8-21 - Procarbazine 75 mg/m2 p.o., Day 29 - Vincristine 1.4 mg/m2 i.v.) followed by radiation therapy (External Beam RT 59.4 Gy (1.8 Gy x 33 fractions, 5 days a week) to MR defined tumor volume).
  Interventions: Drug: lomustine; Drug: procarbazine hydrochloride; Drug: vincristine sulfate; Radiation: radiation therapy

INTERVENTIONS:
Drug: lomustine
  Arms: Intensive pre-treatment chemotherapy and radiation therapy
Drug: procarbazine hydrochloride
  Arms: Intensive pre-treatment chemotherapy and radiation therapy
Drug: vincristine sulfate
  Arms: Intensive pre-treatment chemotherapy and radiation therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy with radiation therapy may kill more tumor cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of radiation therapy with or without chemotherapy in treating patients who have anaplastic oligodendroglioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival and time to tumor progression in patients with unifocal or multifocal, supratentorial, pure or mixed anaplastic oligodendroglioma treated with radiotherapy with or without procarbazine, lomustine, and vincristine (PCV).
* Compare the toxic effects of these 2 regimens in these patients.
* Compare the quality of life and neurologic function of patients treated with these 2 regimens.

OUTLINE: This is a randomized study. Patients are stratified by age (under 50 vs 50 and over), Karnofsky performance status (60-70% vs 80-100%), and tumor grade (moderately vs highly anaplastic). Within 8 weeks after diagnostic surgery, patients are randomized to 1 of 2 treatment arms.

* Arm I: Within 2 weeks after randomization, patients receive oral lomustine on day 1, oral procarbazine on days 8-21, and vincristine IV on days 8 and 29 (PCV). Treatment continues every 6 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Beginning within 6 weeks after day 29 of course 4, patients undergo radiotherapy 5 days a week for 5.6 weeks followed by boost radiotherapy 5 days a week for 1 week.
* Arm II: Within 2 weeks after randomization, patients undergo radiotherapy as in arm I.

Quality of life is assessed at baseline; at time of CT or MRI scans during study; and every 3 months for 1 year, every 4 months for 1 year, every 6 months for 3 years, and then annually thereafter after completion of study therapy.

Patients are followed every 3 months for 1 year, every 4 months for 1 year, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 292 patients (146 per arm) will be accrued for this study within 5.4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven unifocal or multifocal, supratentorial, pure or mixed anaplastic oligodendroglioma

  * Prior suspected or proven low-grade glioma allowed if current histologic proof of pure or mixed anaplastic oligodendroglioma
* Tumor must contain an unequivocal (at least 25%) oligodendroglial element and have 2 or more anaplastic features, 1 of which must be frequent mitoses or endothelial proliferation

  * For mixed tumors, the non-oligodendroglial element must be astrocytic and the oligodendroglial or astroglial component may be anaplastic
* No evidence of spinal drop metastasis or spread to noncontiguous meninges

  * MRI of spine not required for asymptomatic patients and patients not excluded based on pathologic evidence of local meningeal infiltration by underlying tumor
* No tumor that is predominantly located in the posterior fossa (i.e., brainstem or cerebellum)
* No spinal cord tumors

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 150,000/mm^3

Hepatic:

* Bilirubin no greater than 2 times normal
* Serum glutamate oxaloacetate transaminase (SGOT) no greater than 2 times normal
* Alkaline phosphatase no greater than 2 times normal

Renal:

* Creatinine no greater than 1.5 times normal

Pulmonary:

* No chronic lung disease unless diffusion capacity of lung for carbon monoxide (DLCO) is at least 60% predicted

Other:

* No active infection
* No other malignancy within the past 5 years except nonmelanomatous skin cancer or carcinoma in situ of the cervix
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* No concurrent steroids as antiemetics
* Concurrent steroids allowed to control central nervous system (CNS) symptoms due to tumor-associated or radiotherapy-associated cerebral edema

Radiotherapy:

* No prior radiotherapy to brain or head/neck

Surgery:

* Prior surgery allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 1994-07 (Actual); Primary Completion 2005-02 (Actual); Study Completion 2018-05-21 (Actual)

PRIMARY OUTCOMES:
Overall Survival | From randomization to date of death or last follow-up. Analysis occurs after all patients have been potentially followed for 3 years.

SECONDARY OUTCOMES:
Time to tumor progression | From randomization to date of progression or last follow-up. Analysis occurs after all patients have been potentially followed for 3 years.
Frequency of severe (>= Grade 3) toxicities | From randomization to date of death or last follow-up. Analysis occurs after all patients have been potentially followed for 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: J. Gregory Cairncross, MD, Study Chair — London Health Sciences Centre; Steven R. Alberts, MD, Study Chair — Mayo Clinic; Karen L. Fink, MD, PhD, Study Chair — Simmons Cancer Center; Richard M. Hellman, MD, Study Chair — Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center; Normand Laperriere, MD, FRCPC, Study Chair — Princess Margaret Hospital, Canada
Locations (95):
- United States (95):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Carl T. Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Veterans Affairs Medical Center - West Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - OHSU Cancer Institute, Portland, Oregon
  - Veterans Affairs Medical Center - Charleston, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington

REFERENCES:
- [Result] Cairncross JG, Wang M, Shaw EG, et al.: Chemotherapy plus radiotherapy (CT-RT) versus RT alone for patients with anaplastic oligodendroglioma: long-term results of the RTOG 9402 phase III study. [Abstract] J Clin Oncol 30 (Suppl 15): A-2008b, 2012.
- [Result] Wang M, Cairncross G, Shaw E, Jenkins R, Scheithauer B, Brachman D, Buckner J, Fink K, Souhami L, Laperriere N, Mehta M, Curran W; Radiation Therapy Oncology Group (RTOG); North Central Cancer Treatment Group (NCCTG); Southwest Oncology Group (SWOG); National Cancer Institute of Canada Clinical Trials Group (NCIC CTG); Eastern Cooperative Oncology Group (ECOG). Cognition and quality of life after chemotherapy plus radiotherapy (RT) vs. RT for pure and mixed anaplastic oligodendrogliomas: radiation therapy oncology group trial 9402. Int J Radiat Oncol Biol Phys. 2010 Jul 1;77(3):662-9. doi: 10.1016/j.ijrobp.2009.06.004. Epub 2009 Sep 23. PMID 19783377
- [Result] Giannini C, Burger PC, Berkey BA, Cairncross JG, Jenkins RB, Mehta M, Curran WJ, Aldape K. Anaplastic oligodendroglial tumors: refining the correlation among histopathology, 1p 19q deletion and clinical outcome in Intergroup Radiation Therapy Oncology Group Trial 9402. Brain Pathol. 2008 Jul;18(3):360-9. doi: 10.1111/j.1750-3639.2008.00129.x. Epub 2008 Mar 26. PMID 18371182
- [Result] Intergroup Radiation Therapy Oncology Group Trial 9402; Cairncross G, Berkey B, Shaw E, Jenkins R, Scheithauer B, Brachman D, Buckner J, Fink K, Souhami L, Laperierre N, Mehta M, Curran W. Phase III trial of chemotherapy plus radiotherapy compared with radiotherapy alone for pure and mixed anaplastic oligodendroglioma: Intergroup Radiation Therapy Oncology Group Trial 9402. J Clin Oncol. 2006 Jun 20;24(18):2707-14. doi: 10.1200/JCO.2005.04.3414. PMID 16782910
- [Result] Cairncross G, Seiferheld W, Shaw E, et al.: An intergroup randomized controlled clinical trial (RCT) of chemotherapy plus radiation (RT) versus RT alone for pure and mixed anaplastic oligodendrogliomas: initial report of RTOG 94-02. [Abstract] J Clin Oncol 22 (Suppl 14): A-1500, 107s, 2004.
- [Result] Shaw EG, Seiferheld W, Cairncross JG, et al.: Radiation therapy (RT) alone vs intensive procarbazine-CCNU-vincristine (I-PCV) chemotherapy followed by radiation therapy for anaplastic oligodendroglioma (AO) and mixed oligo-astrocytoma (MOA): results of Radiation Therapy Oncology Group (RTOG) - intergroup protocol 94-02. [Abstract] Int J Radiat Oncol Biol Phys 60 (1 Suppl 1): A-57, S163, 2004.
- [Result] Jenkins RB, Curran W, Scott CB, Cairncross G. Pilot evaluation of 1p and 19q deletions in anaplastic oligodendrogliomas collected by a national cooperative cancer treatment group. Am J Clin Oncol. 2001 Oct;24(5):506-8. doi: 10.1097/00000421-200110000-00018. PMID 11586105
- [Derived] Lassman AB, Hoang-Xuan K, Polley MC, Brandes AA, Cairncross JG, Kros JM, Ashby LS, Taphoorn MJB, Souhami L, Dinjens WNM, Laack NN, Kouwenhoven MCM, Fink KL, French PJ, Macdonald DR, Lacombe D, Won M, Gorlia T, Mehta MP, van den Bent MJ. Joint Final Report of EORTC 26951 and RTOG 9402: Phase III Trials With Procarbazine, Lomustine, and Vincristine Chemotherapy for Anaplastic Oligodendroglial Tumors. J Clin Oncol. 2022 Aug 10;40(23):2539-2545. doi: 10.1200/JCO.21.02543. Epub 2022 Jun 22. PMID 35731991
- [Derived] Cairncross G, Wang M, Shaw E, Jenkins R, Brachman D, Buckner J, Fink K, Souhami L, Laperriere N, Curran W, Mehta M. Phase III trial of chemoradiotherapy for anaplastic oligodendroglioma: long-term results of RTOG 9402. J Clin Oncol. 2013 Jan 20;31(3):337-43. doi: 10.1200/JCO.2012.43.2674. Epub 2012 Oct 15. PMID 23071247